CLINICAL TRIAL: NCT07026929
Title: Tracing the Origin and Progression of Parkinson's Disease Through the Neuro-Immune Interactome
Brief Title: Neuro-immune Interactome in Parkinson's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Fox (Michael J.) Foundation for Parkinson's Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2000029032
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- RBD without motor or cognitive dysfunction: Participants with RBD without motor or cognitive dysfunction, normal DaT Scan, no complaints of constipation, normosmic (at no or remote risk for PD)
- RBD and asymmetric: Participants with RBD and asymmetric, reduced signal on DaT scan, symptomatic constipation, or hyposmia with or without minor motor signs of PD (at-risk for PD)
- RBD with PD: Participants with RBD and PD for less than 10 years (10 years from PD diagnosis at the time subject was first identified to be screened for the study)
- PD without RBD: Participants with PD without RBD
- Healthy controls: no RBD, no PD

SUMMARY:
This study will be observational and have a prospective case-control longitudinal design. Eligible subjects with idiopathic REM behavior disorder (RBD), Parkinson's disease with RBD, and healthy controls will be recruited. Subjects will undergo a sleep study to determine eligibility for the study and then in the study will undergo clinical assessments, including cognitive, sensory and motor clinical assessment, dopamine transporter scanning, and smell testing. Eligible subjects will undergo phlebotomy, lumbar puncture, stool and saliva collection, and genome-wide association scans at baseline and then undergo yearly sensory and motor clinical assessment to assess for phenoconversion to neurodegenerative disease.

From blood and CSF samples, investigators will isolate mononuclear cells, and using cell immunologic and single cell genomic procedures, will look for the presence of T cells which autoreact with alpha-synuclein. Investigators will also look for the presence of increased clonality of T cells reflecting increased immune cell activation and the presence of cross reactivity of anti-alpha-synuclein T cells with microbial agents from subject gut stool samples.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether T cell-mediated autoimmunity initiates the neurodegenerative process in PD, and if these early immunological processes converge on classic archetypes of neurodegeneration.

Secondary objectives of this study are to determine to what extent the T cell-mediated autoimmune process initiates in the gut microbiome; and whether or not different PD- related genes or HLA type are associated with the presence of T cell-mediated autoimmunity.

Investigators hypothesize that progression of Parkinson's Disease (PD) pathology is initiated and/or abetted by an autoimmune process involving alpha-synuclein-specific T cell activation triggered by gut microbiome dysbiosis, followed by neuro-immune interactions that establish PD in the brain. Investigators propose to address this hypothesis by integrating neuroimmunology, single cell genomics, mouse models, and microbiome approaches.

ELIGIBILITY:
Inclusion Criteria:

General:

* English Speaking
* Able and willing to provide informed consent

REM behavior disorder:

* Repeated episodes of sleep-related vocalization and/or complex motor behaviors. These behaviors are documented by polysomnography to occur during REM sleep or, based on clinical history of dream enactment, are presumed to occur during REM sleep.
* Polysomnographic recording demonstrates REM sleep without atonia (RWA).
* The disturbance is not better explained by another sleep disorder, mental disorder, medication, or substance abuse.

Parkinson's disease:

* Meets the Movement Disorders Society criteria for Clinically Probable Parkinson's disease.
* Disease duration < 10 years 10 years from PD diagnosis at the time subject was first identified to be screened for the study.

Healthy controls:

* No clinical evidence of Parkinson's disease or RBD.
* Normosmic.

Exclusion Criteria:

General:

* Known immune deficiency disorder.
* Personal history of any neurological disorder, including but not limited to:

Multiple Sclerosis, Alzheimer's disease, Multiple System Atrophy, Progressive Supranuclear Palsy, Amyotrophic Lateral Sclerosis, or repeated head trauma.

* Solid or hematological malignancy other than in-situ carcinoma of the cervix or basal cell carcinoma of the skin unless the subject has no evidence of active disease and has not received treatment, including chemotherapy, immunotherapy or radiation treatment within previous 12 months.
* Known blood clotting disorder (with increased likelihood of bleeding).
* Short Bowel Syndrome, Ileostomy, or colostomy
* History of vagotomy.
* Taking anticoagulant or antiplatet medication (coumadin, heparin, apixaban (Eliquis ®), rivaroxaban (Xalreto®), edoxaban (Lixiana®), or dabigatran (Praxeda®). Low-dose (100 mg/day or less) aspirin is allowed. Taking certain drugs that can interfere with interpretation of DaT scan, such as methylphenidate (Ritalin®), stimulant drugs such as phentermine or ephedrine, certain antidepressants, including mazindol, or radaraxine, benztropine (Cogentin®) within 5 half-lives prior to the date of the scheduled DaT scan. Subjects taking a potentially interfering medication can only be included if the medication is stopped with the concurrence of the subject and the prescribing health care provider. Persons taking bupropion or amphetamine will be asked to hold the medicine on the morning of the scan. They will be able to take the medicine the same day after the scan. Inability to hold bupropion or an amphetamine for the scan, however, will not exclude an individual from participating.
* Receiving chemotherapy agents with ability to affect the immune system, or radiation therapy (within the past 12 months).
* Receiving potent immunosuppressant agents (e.g., anti-TNF, or IL-6 antibodies, JAK/STAT inhibitors, chemotherapy agents such as methotrexate or Cytoxan used to induce immunosuppression), Use of low, maintenance doses of corticosteroids may be permitted, depending on the underlying disease indication.
* Treatment with an experimental agent within 3 months of screening.
* Pregnancy or actively breast feeding.
* Treatment of thyroid disease with radioactive iodine.
* Lidocaine allergy.

Additional Exclusion Criteria for Subjects with diagnosis of PD:

* Meets any of the MDS exclusionary criteria for PD diagnosis. Additional Exclusion Criteria for Subjects with RBD
* An identified secondary cause of RBD.
* Neurodegenerative Disease: Neurological examination must be performed to exclude parkinsonism (according to MDS PD criteria), and clinically evident dementia.
* Secondary RBD, caused by antidepressant medications (antidepressant- triggered RBD can be included provided that diagnosis is documented of antidepressant medications, and patients can be taking antidepressants during the study).
* Diagnosis of narcolepsy. Additional Exclusion Criteria for Healthy Control Subjects
* History of Parkinson's disease in a first-degree blood relative.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from outpatient neurology and sleep medicine clinics and from the community using flyers and social media postings. Subjects in general will be healthy adults seen in an outpatient research setting. There will be no limitation in ability to move or walk as most subjects will be pre-clinical except for Group 4 which will include persons with only minor motor symptoms (which never includes gait disturbance) of PD.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Characterization of of T cells | 2 months
  Number and types of T cells which autoreact to alpha- synuclein in the blood and cerebral spinal fluid (CSF)

SECONDARY OUTCOMES:
Presence of increased clonality of T cells | 2 months
  The presence of increased clonality of T cells reflecting increased immune cell activation will be assessed in Mononuclear cells (PBMCs) and nucleated cells in the CSF isolated and prepared for single cell RNA sequencing.
presence of cross reactivity of anti-alpha- synuclein T cells | 2 months
  Presence of cross reactivity of anti-alpha- synuclein T cells with microbial agents from subject gut stool samples using cells isolated and prepared for single cell RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Cedarbaum, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data not considered PHI and permitted to be released per participants' consent will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the time of publication of the primary manuscript
Access Criteria: Public